CLINICAL TRIAL: NCT00215280
Title: Studies on the Epidemiology and Control of Mansonella Perstans Infection in Uganda
Brief Title: Epidemiology and Control of Mansonella Perstans Infection in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Ministry of Health, Uganda (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MV917090205
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Mansonelliasis; Pruritus; Lymphoedema; Abdominal Pains
Keywords: Mansonella perstans; microfilaraemia; ivermectin; albendazole; Uganda
MeSH Terms: conditions — Mansonelliasis; Pruritus; Lymphedema; Abdominal Pain; Dipetalonema Infections | interventions — Ivermectin; Albendazole

INTERVENTIONS:
Drug: ivermectin and albendazole

SUMMARY:
Mansonella perstans (M. perstans) infection is widespread in Uganda. Knowledge about the epidemiology of this infection, and of the morbidity it induces is poor, and no effective treatment is available. The study aims at providing data on diagnostic, epidemiological, morbidity and treatment aspects of M. perstans infections in Uganda.

DETAILED DESCRIPTION:
Overall objective: to investigate diagnostic, epidemiological and treatment aspects of M. perstans in Uganda with relevance to control

Specific objectives:

1. To establish the pattern of diurnal periodicity of M. perstans microfilaraemia in humans
2. To establish the patterns of M. perstans microfilaraemia and possible clinical manifestations related to this infection in two communities with medium to high endemicity
3. To determine the efficacy of ivermectin alone and the combination of ivermectin and albendazole on M. perstans microfilaraemia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals >= 5 years with or without M. perstans infection

Exclusion Criteria:

* Individuals < 5 years
* Pregnant women

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-11; Study Completion 2006-02

PRIMARY OUTCOMES:
microfilariae periodicity patterns
epidemiology of M. perstans at community level
clinical spectre among infected
reduction in microfilaraemia

SECONDARY OUTCOMES:
treatment effect on clinical manifestations

CONTACTS AND LOCATIONS:
Overall Officials: Asanta M Asio, Msc, Principal Investigator — Ministry of Health, Uganda
Locations (1):
- Luwero, Luwero and Mukono, Luwero and Mukono Districts, Uganda

REFERENCES:
- [Derived] Asio SM, Simonsen PE, Onapa AW. A randomised, double-blind field trial of ivermectin alone and in combination with albendazole for the treatment of Mansonella perstans infections in Uganda. Trans R Soc Trop Med Hyg. 2009 Mar;103(3):274-9. doi: 10.1016/j.trstmh.2008.10.038. Epub 2008 Dec 9. PMID 19081121
- [Derived] Asio SM, Simonsen PE, Onapa AW. Mansonella perstans filariasis in Uganda: patterns of microfilaraemia and clinical manifestations in two endemic communities. Trans R Soc Trop Med Hyg. 2009 Mar;103(3):266-73. doi: 10.1016/j.trstmh.2008.08.007. Epub 2008 Sep 21. PMID 18809192
- See also: Related Info — http://www.dblnet.dk